CLINICAL TRIAL: NCT04591301
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Clinical Study to Assess the Safety, Tolerability and Pharmacokinetics of HEC113995 PA•H2O Tablets in Healthy Subjects
Brief Title: The Safety, Tolerability, and Pharmacokinetics Study of HEC113995 PA•H2O Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC113995PA•H2O-P-01/CRC-C1910
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- HEC113995 PA•H2O 2.5mg (Experimental): Healthy subjects are given HEC113995 PA•H2O 2.5 mg in a single dose.
  Interventions: Drug: HEC113995 PA•H2O tablets
- HEC113995 PA•H2O 5mg (Active Comparator): Healthy subjects are given HEC113995 PA•H2O 5 mg in a single dose.
  Interventions: Drug: HEC113995 PA•H2O tablets
- HEC113995 PA•H2O 10mg (Active Comparator): Healthy subjects are given HEC113995 PA•H2O 10 mg in a single dose.
  Interventions: Drug: HEC113995 PA•H2O tablets
- HEC113995 PA•H2O 20mg (Active Comparator): Healthy subjects are given HEC113995 PA•H2O 20 mg in a single dose.
  Interventions: Drug: HEC113995 PA•H2O tablets
- HEC113995 PA•H2O 40mg (Active Comparator): Healthy subjects are given HEC113995 PA•H2O 40 mg in a single dose.
  Interventions: Drug: HEC113995 PA•H2O tablets
- HEC113995 PA•H2O 60mg (Active Comparator): Healthy subjects are given HEC113995 PA•H2O 60 mg in a single dose.
  Interventions: Drug: HEC113995 PA•H2O tablets
- HEC113995 PA•H2O 80mg (Active Comparator): Healthy subjects are given HEC113995 PA•H2O 80 mg in a single dose.
  Interventions: Drug: HEC113995 PA•H2O tablets
- placebo (Placebo Comparator): Healthy subjects are given placebo in a single dose.
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: HEC113995 PA•H2O tablets — Each dose of HEC113995 PA•H2O tablets will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  Arms: HEC113995 PA•H2O 10mg; HEC113995 PA•H2O 2.5mg; HEC113995 PA•H2O 20mg; HEC113995 PA•H2O 40mg; HEC113995 PA•H2O 5mg; HEC113995 PA•H2O 60mg; HEC113995 PA•H2O 80mg
Drug: Placebo tablets — Placebo tablets will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  Arms: placebo

SUMMARY:
The Safety, Tolerability and Pharmacokinetics Study of HEC113995 PA•H2O Tablets in Healthy Male and Female Subjects

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who are willing and are able to provide a written informed consent to participate in the study.
* 2. Without Plan for pregnancy or pregnant within 3 months after enrollment throughout the trial.
* 3. Subjects aged between 18 and 45 (both inclusive) years old.
* 4. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥18 and ≤28 kg/m2 at screening.
* 5. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* 1.Subjects with serum creatinine, ALT and AST levels ≥1.5 times of the upper limit of normal value at screening.
* 2.Subjects with a positive serology for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and/or TP antibodies at screening.
* 3. Subjects with history of digestive system,urinary system, liver,central nervous system, blood system, endocrine system,respiratory system,immune system,cardiovascular system,and/or malignant tumor or others medical conditions (such as history of mental illness, etc.) that are not suitable for clinical trial participation;Subjects with history of epilepsy, bipolar disorder/mania, high intraocular pressure, or acute angular-closure glaucoma.
* 4. Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s)# anaphylaxis physique.
* 5. Use of any prescription or non-prescription medications within 14 days prior to initial dosing#Use of any medications known to inhibit or induce cytochrome P enzyme drug metabolism within 28 days prior to initial dosing.
* 6. Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
* 7. Positive results from urine drug screen test.
* 8. History of alcoholism or drink regularly within 3 months prior to the study(defined as Alcohol consumption of > 21 units/week), or positive results from alcohol breath test.
* 9.Regular smoking of more than 10 cigarettes per day within 3 months before administration of study drug, or inability to refrain from smoking during the course of the study.
* 10. Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
* 11. Subjects who plan to receive or have had organ transplants.
* 12. Subjects who participated in another clinical trial within 3 months prior to initial dosing.
* 13. Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of HEC113995 PA•H2O by Assessment of the Number of Adverse Events (AEs) Following Administration in Single Ascending Dose | up to 7 days
  To investigate the safety and tolerability of HEC113995 PA•H2O by assessment of AEs (non-serious and serious) following administration in SAD

SECONDARY OUTCOMES:
PK parameters - AUC0-∞ | up to 144 hours
  area under the concentration versus time curve (AUC) from time zero to infinity
PK parameters - Cmax | up to 144 hours
  Geometric Mean of Maximum Observed Plasma Concentration of HEC113995 PA•H2O
PK parameters -tmax | up to 144 hours
  time to peak
PK parameters -t½ | up to 144 hours
  apparent terminal elimination half-life
PK parameters -Vz/F | up to 144 hours
  apparent volume of distribution
PK parameters - MRT | up to 144 hours
  the Mean Residence Time
PK parameters -CL/F | up to 144 hours
  the Apparent Clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China